CLINICAL TRIAL: NCT02486445
Title: Rivaroxaban for Scheduled Work-up of Patients With Suspected Deep Venous Thrombosis
Brief Title: Rivaroxaban for Scheduled Work-up of DVT - The Ri-Schedule Study
Acronym: Ri-Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3304
Record Dates: First submitted 2015-02-25; First posted 2015-07-01 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2017-09

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep venous thrombosis; Rivaroxaban
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivaroxaban (Experimental): Rivaroxaban 15 mg every 12 hours until the completion of the diagnostic work-up, which should not exceed 24 hours.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15 mg every 12 hours until the completion of the diagnostic work-up, which should not exceed 24 hours (maximum 2 tablets)
  Other Names: Xarelto

SUMMARY:
This prospective outcome study is designed to assess the safety of rivaroxaban in the pre-diagnosis phase of DVT.

DETAILED DESCRIPTION:
This prospective outcome study is designed to assess the safety of rivaroxaban in the pre-diagnosis phase of DVT.

International guidelines suggest the use of low molecular weight heparin (LMWH) if the diagnostic process is expected to be delayed for more than 4 hours.

Rivaroxaban is a new DOAC that in clinical trials has proven to be non-inferior to LMWH and warfarin for the treatment of DVT with the added benefit of causing less major bleeding.

Because of its rapid onset of action and oral administration, rivaroxaban could be used instead of LMWH in the pre-diagnosis phase pending the results of the diagnostic test. However, the safety of a such proposed indication has to be proven before it can be adopted in clinical practice.

This study aims to determine the safety and feasibility of pre-diagnostic treatment with rivaroxaban. The primary outcome of this study "safety" is a composite endpoint of serious bleedings encountered within 48 hours after administration of rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive outpatients referred to ER because of suspected DVT
* 18 years of age
* Signed informed consent

Exclusion Criteria:

1- refuse to consent

Patients with the criteria below will not be eligible for scheduled work-up:

1. Duration of the diagnostic work-up is expected to last < 2 hours
2. Presence of active cancer or receiving chemotherapy for cancer
3. Suspicion of coexisting clinical PE
4. Suspicion of active bleeding (gastrointestinal bleeding or muscle hematoma)
5. Signs of threatened circulation or having intractable pain in the lower extremity or may be considered as candidate for thrombolytic treatment
6. Physician does not consider it safe to discharge the patient
7. Presence of logistic factors that may hinder a scheduled work-up
8. Presence of co-morbid conditions that require hospital admission
9. Patient prefers not to be discharged before diagnosis is completed
10. Glomerular Filtration Rate < 45 ml/min
11. Presence of contraindications to rivaroxaban including;

    * Lesion or condition, if considered to be a significant risk for major bleeding e.g current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities
    * Concomitant treatment with any other anticoagulants e.g. unfractionated heparin (UFH), low molecular weight heparins (enoxaparin, dalteparin, etc.), heparin derivatives (fondaparinux, etc.), oral anticoagulants (warfarin, dabigatran etexilate, apixaban etc.)
    * Hepatic disease associated with coagulopathy and clinically relevant bleeding risk including cirrhotic patients with Child Pugh B and C.
    * Pregnancy/positive pregnancy test and breastfeeding (see section 4.6)

11. Hb < 11 g/dl 12. Presence of drug interaction with rivaroxaban including concomitant systemic treatment with azole-antimycotics (such as ketoconazole, itraconazole, voriconazole and posaconazole) or HIV protease inhibitors (e.g. ritonavir), acetylsalicylic acid at a dose higher than 160 mg or platelet aggregation inhibitors

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of serious bleedings and/or death related to bleeding | Until 48 hours after last tablet
  Serious bleedings and/or death related to bleeding encountered within 48 hours after the last rivaroxaban tablet was ingested in patients in whom DVT was excluded or until the ingestion of first tablet of oral anticoagulation or application of IV/SC heparin in those in whom DVT is confirmed.

SECONDARY OUTCOMES:
Feasability rate | 12 hours
  Assessed by the proportion of patients who can be managed by a scheduled work-up
Failure rate | until 48 hours after last tablet
  Worsening in pre-existing complaints or developement of signs/symptoms of pulmonary embolism
90-day outcome | 90 days
  The 90-day outcome of the applied diagnostic strategy using Wells pre-test clinical probability, D-dimer and compression ultrasounography and safety of coagulation

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghanima, PhD, Study Director — Ostfold Hospital Trust; Nezar Raouf, Principal Investigator — Ostfold Hopital Trust; Kristin Utne, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Ostfold Hospital Trust, Fredrikstad, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Derived] Mohamad H, Jorgensen CT, Ghanima W, Tavoly M, Fronas SG. Clinical use and safety of empiric anticoagulation during diagnostic work-up for deep vein thrombosis. Hematology. 2025 Dec;30(1):2573586. doi: 10.1080/16078454.2025.2573586. Epub 2025 Oct 20. PMID 41116683
- [Derived] Fronas SG, Jorgensen CT, Dahm AEA, Wik HS, Gleditsch J, Raouf N, Holst R, Klok FA, Ghanima W. Safety of a strategy combining D-dimer testing and whole-leg ultrasonography to rule out deep vein thrombosis. Blood Adv. 2020 Oct 27;4(20):5002-5010. doi: 10.1182/bloodadvances.2020002173. PMID 33057634
- [Derived] Fronas SG, Dahm AEA, Wik HS, Jorgensen CT, Gleditsch J, Raouf N, Holst R, Klok FA, Ghanima W. Safety and feasibility of rivaroxaban in deferred workup of patients with suspected deep vein thrombosis. Blood Adv. 2020 Jun 9;4(11):2468-2476. doi: 10.1182/bloodadvances.2020001556. PMID 32502267